CLINICAL TRIAL: NCT02573558
Title: Prevalence of Postoperative Delirium According to the Use of Dexmedetomidine or Propofol in Elderly Patients Undergoing Orthopedic Surgery: Retrospective Study
Brief Title: Intraoperative Sedation and Postoperative Delirium
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Associate Professor, Seoul National University Bundang Hospital
Other Study IDs: B-1510/318-104
Record Dates: First submitted 2015-10-06; First posted 2015-10-12 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Orthopedics
MeSH Terms: interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- DEX: patients who received dexmedetomidine during the operation
  Interventions: Drug: Dexmedetomidine
- PPF: patients who received propofol during the operation
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Dexmedetomidine
  Groups: DEX
Drug: Propofol
  Groups: PPF

SUMMARY:
Delirium are common after orthopedic surgery in the elderly and are directly associated with loss of independence, reduction in the quality of life and increased mortality. The cause of postoperative delirium still remains unclear and may be multifactorial. The aim of this retrospective study is to examine prevalence of postoperative delirium according to the use of dexmedetomidine or propofol in elderly patients undergoing orthopedic surgery under regional anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent orthopedic surgery under regional anesthesia
* age of 65 years or greater

Exclusion Criteria:

* General anesthesia
* age < 65 years
* central nervous system disease, including dementia and Parkinson's disease
* Patients who were not received sedation with propofol or dexmedetomidine during the operation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients who underwent orthopedic surgery under regional anesthesia, and age of 65 years or greater
Sampling Method: Probability Sample
Enrollment: 855 (Actual)
Dates: Start 2015-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
delirium | within 7 day postoperatively

SECONDARY OUTCOMES:
Wound infection | within 7 day postoperatively
Pulmonary thromboembolism | within 7 day postoperatively
Hospital stay | through study completion, an average of 7days

OTHER OUTCOMES:
Myocardial ischemia | within 7 day postoperatively
Renal failure | within 7 day postoperatively
Hepatic failure | within 7 day postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea